CLINICAL TRIAL: NCT01842217
Title: Validation of [18F]FES for Imaging of Brain Estrogen Receptors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL41 608.042.12
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Psychiatric/Mood Disorder | Patient; Estrogen Receptor Levels; Premenopausal; Postmenopausal
Keywords: 18F-FES PET; Nuclear Medicine; Premenopausal; Postmenopausal; Estrogen receptor; Anxiety; Depression; Cognition
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Premenopausal women (Other): healthy female subjects: premenopausal
  Interventions: Procedure: FES-PET
- Postmenopausal women (Other): healthy female subjects: postmenopausal
  Interventions: Procedure: FES-PET

INTERVENTIONS:
Procedure: FES-PET

SUMMARY:
Validation of [18F]-FES for imaging of estrogen receptors in the brain

The primary objective of the study is to determine if [18F]-FES Positron Emission Tomography (PET) can be used to quantify the estrogen receptor expression in the human brain.

DETAILED DESCRIPTION:
Estrogens are the primary female sex hormones that play a major role in the development and maintenance of secondary sexual functions. In addition, estrogens play an important role in cardiovascular, musculoskeletal, immunological, bone development and central nervous system processes. Actions of estrogens are mediated by a group of specialized receptors, known as estrogen receptors. Estrogens were found to be neuroprotective and may thus protect against development of neurodegenerative disorders like Alzheimer's disease, Parkinson's disease and multiple sclerosis. In addition, estrogens may also play an important role in psychiatric disorders, like depression. To improve our understanding of the action of estrogens in the brain, it is important to study the expression of estrogen receptors in the brain. Positron emission tomography (PET) is the most suitable technique for non-invasive imaging of brain receptors. [18F]FES is a PET tracer that is regularly used in the UMCG to image the estrogen receptor expression in breast cancer patients, but has never been used for quantitative imaging of brain estrogen receptors. Quantification of the expression of brain receptors by PET usually requires arterial blood sampling to obtain the plasma input function of the tracer. Arterial blood sampling causes discomfort to the patient and therefore can be an obstacle especially in longitudinal studies. The aim of this study is therefore to investigate whether [18F]FES PET imaging for quantification of estrogen receptors in the human brain is feasible without arterial blood sampling, using a reference tissue model (SRTM) or an image derived input function (IDIF), so the discomfort associated with arterial blood sampling can be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years
* For postmenopausal women: at least 1 year after menopause
* For premenopausal women: a regular menstruation
* Signed written informed consent

Exclusion Criteria:

* Use of estrogen receptor ligands, such as tamoxifen or fulvestrant
* History of ER-positive malignancies or breast cancer
* Use of any contraceptive drugs (pill, injections or implanted)
* For postmenopausal women: (history of) estrogen replacement therapy
* Pregnancy
* History of removal of the ovaries and/or the uterus
* Current systemic diseases
* Major metabolic diseases (e.g. diabetes, hyper- or hypothyroidism)
* Somatic, organic or neurological disorders
* Recent participation in a scientific research study (<1 year) involving radiation
* Claustrophobia
* Presence of materials in the body that can be magnetized, like: pacemaker, metallic implants/prostheses, metal fragments, shunts, artificial heart valves, vascular clips, fixed hearing aid, tattoos containing metal, hair implants, artificial dentures

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quantification of estrogen receptors in the human brain | 1 year
  The primary objective of the study is to validate the use of a reference tissue model and an image derived input function for the quantification of ERs in the human brain, by [18F]FES PET, using pharmacokinetic modelling with arterial sampling as golden standard

SECONDARY OUTCOMES:
Evalution of the levels of circulating estradiol in two patient cohorts and to evaluate the imaging technique | 1 year
  1. To evaluate the effect of the levels of circulating estradiol on quantification of ERs in the human brain, by comparing premenopausal women with postmenopausal women.
  2. To investigate whether PET acquisition time can be shortened to reduce the subjects discomfort, as the current protocol requires the patient to be scanned for 90 min.

CONTACTS AND LOCATIONS:
Overall Officials: Andor Glaudemans, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands